CLINICAL TRIAL: NCT03221231
Title: N-acetylcysteine for the Treatment of Cannabis Dependence: Working Mechanisms
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 131115
Record Dates: First submitted 2017-06-19; First posted 2017-07-18 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Cannabis Use Disorder; Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Acetylcysteine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- N-acetylcysteine (Experimental)
  Interventions: Drug: N-acetylcysteine; Other: Magnetic Resonance Imaging; Other: Neurocognitive measures; Other: Neuro-inflammatory measures
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet; Other: Magnetic Resonance Imaging; Other: Neurocognitive measures; Other: Neuro-inflammatory measures
- Healthy controls (Active Comparator)
  Interventions: Other: Magnetic Resonance Imaging; Other: Neurocognitive measures; Other: Neuro-inflammatory measures

INTERVENTIONS:
Drug: N-acetylcysteine — 1200 mg/day, twice daily, N-acetylcysteine
  Arms: N-acetylcysteine
Drug: Placebo Oral Tablet — twice daily, placebo
  Arms: Placebo
Other: Magnetic Resonance Imaging
Other: Neurocognitive measures
Other: Neuro-inflammatory measures

SUMMARY:
This study investigates the effects of repeated NAC administration on glutamate concentrations in the anterior cingulate cortex (ACC), on neurocognitive functioning, and on neuro-inflammatory parameters in adult cannabis-dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV diagnosis of cannabis dependence, >1 week detoxified and abstinent;
* Able to provide written informed consent and to comply with study procedures.
* Dutch speaking (Dutch as primary language).

Exclusion Criteria:

* Currently dependent on any substance other than cannabis, alcohol or nicotine;
* History of any major internal disease (including diabetes, cardiovascular disease, lung disease, liver or kidney disease);
* An active or any history of neurological disorder, including but not limited to seizure disorder, epilepsy, stroke, neurological disease, cognitive impairment, head trauma with prolonged loss of consciousness (>10 minutes), or migraine headaches;
* An active or a history of a psychiatric disorder including, but not limited to, depression, schizophrenia, bipolar disorder, anxiety, or other psychiatric disorders;
* Asthma;
* Known hypersensitivity or allergy to n-acetylcysteine, or receiving chronic therapy with medication that could interact adversely with n-acetylcysteine within 30 days prior to randomization (i.e., nitroglycerin, ACE inhibitors or antihypertensive drugs, anti-coagulants);
* Exclusion criteria for MRI: having metal in the body and/or having claustrophobia

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-05-15 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Brain glutamate concentrations | at study end (2 weeks after study start)
  Glutamate concentrations in the anterior cingulate cortex (ACC)

SECONDARY OUTCOMES:
Motor impulsivity | at study end (2 weeks after study start)
  Stop Signal Reaction Time (SSRT) on the Stop Signal Task
Cognitive impulsivity | at study end (2 weeks after study start)
  Indifference point measured by a Monetary Delayed Discounting Task
Attentional Bias | at study end (2 weeks after study start)
  Difference in response time for incongruent-congruent stimuli on a Stroop task
Neuro-inflammation | at study end (2 weeks after study start)
  Concentration of interleukin in blood

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Brussels, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided